CLINICAL TRIAL: NCT06739603
Title: Impact of Renal Function Availability to Community Pharmacist for Dispensing Direct Oral Anticoagulant in Ambulatory Patients on Bleeding Occurrence
Acronym: Hemorrag-IR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023_RIPH_007_Hemorrag-Ir
Record Dates: First submitted 2024-12-12; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: AOD Prescription
Keywords: community pharmacist; AOD; renal function; bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : pharmaceutical analysis of the prescription of Direct Oral Anticoagulant (Experimental): community pharmacist makes every effort to obtain the patient's renal function in order to carry out a pharmaceutical analysis of the prescription of Direct Oral Anticoagulant
  Interventions: Other: pharmaceutical analysis
- Group 2 : control group (No Intervention): No intervention (the community pharmacist takes no additional action to improve the patient's renal function)

INTERVENTIONS:
Other: pharmaceutical analysis — pharmaceutical analysis
  Arms: Group 1 : pharmaceutical analysis of the prescription of Direct Oral Anticoagulant

SUMMARY:
The use of direct oral anticoagulants (AODs) in the prevention and treatment of thromboembolic diseases is increasing, with a favorable benefit/risk balance and improved quality of life for patients. However, anticoagulants are still associated with a risk of bleeding, making them one of the drugs most likely to cause adverse events and serious adverse events. Certain clinical situations are particularly at risk of bleeding with AODs, notably renal failure (even moderate) and age over 75, due to the predominant renal elimination of these drugs. Prescription and monitoring of AOD treatment are conditional on monitoring of renal function and, if necessary, appropriate dosage adjustments.

Community pharmacists dispense AODs on a daily basis, following pharmaceutical analysis. Good dispensing practice recommends that community pharmacists have access to biological data. Studies have suggested that access to renal function enables community pharmacists to carry out targeted and appropriate interventions. This expected clinical pharmaceutical expertise is conditional on access to this biological data. In practice, community pharmacists are not systematically aware of this renal function, and are therefore unable to carry out a pharmaceutical intervention if necessary. Initiatives implemented by general practitioners seem to be emerging (systematic addition of the renal to the medical prescription), but these practices do not currently guarantee systematic access to this data. A strong argument in favor of systematically making the renal available to community pharmacists would be to demonstrate that access to this biological data reduces the occurrence of adverse events linked to AODs.

DETAILED DESCRIPTION:
The main objective is to study the benefit of access to the patient's renal function by the dispensing pharmacist when dispensing an AOD (first prescription or renewal) on the occurrence of clinically significant bleeding at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* with a prescription for an AOD (first prescription or renewal),
* whatever the indication of the AOD treatment,
* coming to one of the study's partner pharmacies for dispensing,
* adults,
* agreeing to take part in the study (by signing the informed consent form).

Exclusion Criteria:

* prescribed another class of anticoagulant,
* minors,
* pregnant and breast-feeding women
* who do not understand French
* protected by law (guardianship, curatorship, safeguard of justice),
* refusing to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1920 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
clinically significant bleeding at 3 months | Month 3
  Bleeding requiring unscheduled consultation with general practitioner or specialist, regardless of the type of treatment required (therapeutic abstention, medical management with or without hospitalization, surgical management) and regardless of the type of AOD's treatment management (no change, change or discontinuation)

SECONDARY OUTCOMES:
clinically significant bleeding at 6 months | Month 6
  Bleeding requiring unscheduled consultation with general practitioner or specialist, regardless of the type of treatment required (therapeutic abstention, medical management with or without hospitalization, surgical management) and regardless of the type of AOD's treatment management (no change, change or discontinuation)
major bleeding at 3 months | Month 3
  Bleeding requiring hospitalization or bleeding from a critical organ (intracerebral, intraocular, tamponade, …)
major bleeding at 6 months | Month 6
  Bleeding requiring hospitalization or bleeding from a critical organ (intracerebral, intraocular, tamponade, …)

IPD SHARING:
Plan to Share IPD: Undecided